CLINICAL TRIAL: NCT06795503
Title: Non-Inferiority Study on MRNA-lncRNA Model in Low-Risk Triple-Negative Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2407299-27
Record Dates: First submitted 2024-10-04; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Epirubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Docetaxel plus cyclophosphamide
  Interventions: Drug: Docetaxel plus cyclophosphamide
- Control group (Active Comparator): Epirubicin, cyclophosphamide followed by paclitaxel
  Interventions: Drug: Epirubicin, cyclophosphamide plus paclitaxel

INTERVENTIONS:
Drug: Docetaxel plus cyclophosphamide — Docetaxel (T) at a dose of 75 mg/m² was administered intravenously on Day 1 of each cycle, and Cyclophosphamide (C) at a dose of 600 mg/m² was administered intravenously on Day 1 of each cycle as well.
  Arms: Experimental group
Drug: Epirubicin, cyclophosphamide plus paclitaxel — Patients in the control group received the EC-P regimen chemotherapy, with a cycle length of 21 days, for a total of 8 cycles. The specific treatment was as follows: Epirubicin (E) at a dose of 90 mg/m² and Cyclophosphamide (C) at a dose of 600 mg/m² were administered intravenously on Day 1 of each cycle for the first 4 cycles. This was followed by Paclitaxel (P) at a dose of 80 mg/m², administered intravenously on Days 1, 8, and 15 of each cycle for the subsequent 4 cycles.
  Arms: Control group

SUMMARY:
To compare the efficacy and safety of different adjuvant chemotherapy regimens for low-risk triple-negative breast cancer patients predicted by mRNA-lncRNA model

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged ≥18 and ≤70 years.
2. ECOG performance status of 0 to 1.
3. Histologically confirmed invasive triple-negative breast cancer (TNBC), defined as breast cancer with estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2) all determined to be negative by pathological testing. Specifically, ER-negative: IHC <1%, PR-negative: IHC <1%, HER2-negative: IHC -/+ or IHC++ but FISH/CISH negative. Tissue samples must be verified by the central lead institution as low-risk according to the mRNA-lncRNA model.
4. Postoperative early-stage breast cancer patients who have undergone radical surgery, with pathological TNM staging of pT1c-3N0-3M0.
5. Normal major organ function, meeting the following criteria: ① Hematological examination standards: HB ≥ 90g/L (no blood transfusion within the last 14 days); ANC ≥ 1.5×10⁹/L; PLT ≥ 75×10⁹/L; ② Biochemical examination standards: TBIL ≤ 1.5×ULN (upper limit of normal); ALT and AST ≤ 3×ULN; Serum Cr ≤ 1×ULN, and creatinine clearance rate > 50ml/min (Cockcroft-Gault formula).
6. Women of childbearing potential must use medically approved contraception during the study treatment period and for at least 3 months after the last dose of the study drug.
7. Participants must voluntarily join the study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up procedures.

Exclusion Criteria:

1. Patients who have received neoadjuvant treatment, including chemotherapy, targeted therapy, radiotherapy, or endocrine therapy.
2. Bilateral breast cancer.
3. Metastasis at any site.
4. Any >T4 lesions (UICC1987) (involving skin invasion, tumor fixation, or inflammatory breast cancer).
5. History of clinically significant or uncontrolled heart disease, including congestive heart failure, angina, myocardial infarction within the past 6 months, or ventricular arrhythmias.
6. History of other malignancies within the past 5 years, except for cured in situ cervical cancer, basal cell carcinoma, or squamous cell carcinoma of the skin.
7. Pregnant or breastfeeding women, or women of childbearing potential who are unable to use effective contraception.
8. Patients concurrently participating in other clinical trials.
9. Severe or uncontrolled infections.
10. Known active HBV or HCV infection, or HBV DNA ≥ 500, or chronic infection with abnormal liver function.
11. History of substance abuse that cannot be quit or any psychiatric disorders.
12. Patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1462 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival (iDFS) | Five years
  Invasive disease-free survival (iDFS) is the time after initial cancer treatment during which a patient remains free from invasive cancer recurrence. It's an important measure in clinical trials to assess how well treatments prevent the return of cancer or the development of new invasive cancers after the primary treatment has been completed.

SECONDARY OUTCOMES:
Distant recurrence-free survival (DRFS) | Five years
  Distant recurrence-free survival (DRFS): This refers to the length of time after primary cancer treatment during which a patient does not experience cancer recurrence in distant organs or sites. DRFS is commonly used to evaluate the effectiveness of treatments in preventing metastasis or the spread of cancer to distant parts of the body.
Overall survival (OS) | Five years
  Overall survival (OS): OS is the time from the start of treatment or diagnosis until death from any cause. It is the most direct and important endpoint in clinical trials, measuring the effectiveness of a treatment in extending a patient's life.
Safety according to CTCAE v5.0 (Common Terminology Criteria for Adverse Events, version 5.0) | Five years
  Safety according to CTCAE v5.0: This refers to the assessment of adverse events or side effects of treatment based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. It provides a standardized way to evaluate and report the severity and frequency of treatment-related toxicities to ensure patient safety.